CLINICAL TRIAL: NCT00470275
Title: Phase II Trial of Intermediate-Dose Cytarabine to Modulate EWS/FLI for Children and Young Adults With Recurrent or Refractory Ewing Sarcoma
Brief Title: Cytarabine in Treating Young Patients With Recurrent or Refractory Ewing's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEWS0621; CDR0000542650 (Other: Clinical Trials.gov); COG-AEWS0621 (Other: Children's Oncology Group)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Sarcoma
Keywords: recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cytarbine (Experimental): Cytarabine IV every 12 hours days 1-5 of 21 day cycle. Response evaluation after 6 cycles of therapy.
  Interventions: Drug: cytarabine

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: cytosine arabinoside; Ara-C; Cytosar; NSC #063878

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well cytarabine works in treating young patients with recurrent or refractory Ewing's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in younger patients with recurrent or refractory Ewing's sarcoma treated with cytarabine.

OUTLINE: This is a multicenter study.

Patients receive cytarabine IV over 2 hours twice daily on days 1-5. Treatment repeats every 21 days for up to 11 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Ewing's sarcoma or primitive neuroectodermal tumor (PNET)
* Disease that has recurred or not responded despite prior therapy

  * Has declined enrollment on or is not eligible for clinical trial COG-AEWS0521
* Must have at least one site of measurable disease involving lung or soft tissue as documented by CT scan and/or MRI
* No disease limited to bone

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (for patients > 16 years of age) OR Lansky PS 50-100% (for patients ≤ 16 years of age)
* Life expectancy ≥ 8 weeks
* ANC ≥ 750/mm^3
* Platelet count ≥ 75,000/mm^3 (50,000/mm^3 if documented bone marrow metastatic disease) (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (red blood cell transfusions allowed)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age and < 2.0 mg/dL
* ALT ≤ 2.5 times ULN
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR creatinine meeting the following criteria:

  * ≤ 0.4 mg/dL (1 month to < 6 months of age)
  * ≤ 0.5 mg/dL (6 months to < 1 year of age)
  * ≤ 0.6 mg/dL (1 to < 2 years of age)
  * ≤ 0.8 mg/dL (2 to < 6 years of age)
  * ≤ 1.0 mg/dL (6 to < 10 years of age)
  * ≤ 1.2 mg/dL (10 to < 13 years of age)
  * ≤ 1.4 mg/dL (≥ 13 years of age) (female)
  * ≤ 1.5 mg/dL (13 to < 16 years of age) (male)
  * ≤ 1.7 mg/dL (≥ 16 years of age) (male)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection, including systemic fungal infections requiring ongoing antifungal therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior tumor-directed therapy
* At least 7 days since prior biologic therapy or immunotherapy
* At least 1 week since prior hematopoietic growth factors (2 weeks for pegfilgrastim)
* At least 2 weeks since prior myelosuppressive chemotherapy
* At least 2 weeks since prior local palliative (small-port) radiotherapy
* At least 6 weeks since prior substantial bone marrow radiotherapy
* At least 6 months since prior radiotherapy to ≥ 50% of the pelvis
* At least 6 months since prior autologous stem cell transplantation
* No prior allogeneic stem cell transplantation
* No prior cytarabine
* No other concurrent investigational agents, including chemotherapy, immunotherapy, or biologic therapy
* No other concurrent anticancer chemotherapy or immunomodulating agents

  * Concurrent corticosteroids allowed
* No concurrent intrathecal chemotherapy
* Concurrent radiotherapy to localized painful lesions allowed provided at least one measurable lesion is not irradiated (no irradiated lesion may be used to assess tumor response)

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Stegmaier, MD, Study Chair — Dana-Farber Cancer Institute; Holcombe E. Grier, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (73):
- United States (63):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - Saint Louis, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (8):
  - University of Alberta Hospital, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Result] DuBois SG, Krailo MD, Lessnick SL, Smith R, Chen Z, Marina N, Grier HE, Stegmaier K; Children's Oncology Group. Phase II study of intermediate-dose cytarabine in patients with relapsed or refractory Ewing sarcoma: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2009 Mar;52(3):324-7. doi: 10.1002/pbc.21822. PMID 18989890

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytarbine
Started | 10
Completed | 0
Not Completed | 10
Not completed — Death | 1
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cytarbine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 8
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Any patient who is enrolled and receives at least one dose of cytarabine will be considered evaluable for response if (1) the patient demonstrates progressive disease while on protocol therapy or (2) the patient is observed on protocol therapy for at least one cycle. Patients who achieve a complete or partial response according to the RECIST (Response Evaluation Criteria In Solid Tumors) criteria will be considered responders for the study design. All other patients who are evaluable for response will be considered non-responders for the study.
Time Frame: the first six cycles of study chemotherapy (126 days)
Measure: Number; unit: participants
Groups:
- Cytarabine: Cytarabine IV every 12 hours days 1-5 of 21 day cycle. Response evaluation after 6 cycles of therapy.
Arm/Group | Cytarabine
Number analyzed (Participants) | 10
participants
  Non Responder | 10
  Responder | 0

ADVERSE EVENTS:
Arm/Group | Cytarabine
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytarabine (N=10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytarabine (N=10)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 5
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Conjunctivitis infective (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Eye disorders - Other (Eye disorders) | 1
Facial pain (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Fever (General disorders) | 2
Headache (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Infections and infestations - Other (Infections and infestations) | 5
Lymphocyte count decreased (Investigations) | 3
Nausea (Gastrointestinal disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 8
Non-cardiac chest pain (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Photophobia (Eye disorders) | 1
Platelet count decreased (Investigations) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
White blood cell decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.